CLINICAL TRIAL: NCT06061341
Title: Usage of TruGraf Liver Gene Expression to Identify Subclinical Rejection as Well as Adjust Immunosuppression Medications in Liver Transplant Recipients Due to Autoimmune Disease
Brief Title: TruGraf Liver Gene Expression Serial Test
Status: Enrolling by invitation | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Transplant Genomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 202307175
Record Dates: First submitted 2023-09-20; First posted 2023-09-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Liver Disease; Autoimmune Hepatitis; Primary Sclerosing Cholangitis; Primary Biliary Cirrhosis
MeSH Terms: conditions — Hepatitis, Autoimmune; Cholangitis, Sclerosing; Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TruGraf: Group who will have immunosuppression (IS) assessed utilizing TruGraf Liver Gene Expression test to serially monitor liver transplant recipients with autoimmune disease and alter IS based on these results.
  Interventions: Diagnostic Test: TruGraf®
- Matched historical control group: Group who will have immunosupression (IS) assessed utilizing traditional clinical parameters for IS management.

INTERVENTIONS:
Diagnostic Test: TruGraf® — TruGraf® is a non-invasive blood-based test to assist the clinician in lowering immunosuppression in liver transplant patients. It is the first and only blood-based test that offers biomarker guidance to aid physicians in minimizing immunosuppression in transplant recipients.
  Groups: TruGraf

SUMMARY:
This is an Investigator Initiated, single center, non-randomized, single arm study utilizing TruGraf liver gene expression serial testing in patients with autoimmune liver diseases (AIH, PSC, PBC) monthly for the first 6 months after transplant to help inform immunosuppression (IS) optimization. Approximately 20 patients will be enrolled in the study. Study outcomes will include 1-year graft survival, 1 year BPAR and clinically treated rejection rates, number of changes to IS based on the results of Trugraf, eGFR and immune mediated issues.

TruGraf®, (Transplant Genomics, Inc., a member of Eurofins Transplant Diagnostics) is a non-invasive blood-based test to assist the clinician in lowering immunosuppression in liver transplant patients. It is the first and only blood-based test that offers biomarker guidance to aid physicians in minimizing immunosuppression in transplant recipients. Unfortunately, achieving the tight control of therapeutic levels of immunosuppression that is required to maintain the balance between "too much" and "too little" can be difficult. TruGraf liver can help clinicians confirm immune "quiescence" prior to, as well as following, immunosuppression reduction in patients with stable graft function, minimizing the risk of overt graft injury due to rejection.

The clinical context of use for TruGraf is to provide reassurance to the clinician who is contemplating a preemptive reduction in IS therapy that a patient's immune status is "quiescent" thus reducing the risk of triggering acute rejection with that IS reduction. Having the ability to assess whether the patient's immune status is "quiescent" or activated when considering an increase or decrease in IS therapy allows the clinician greater confidence in decision making.

DETAILED DESCRIPTION:
Study Abstract Following liver transplantation, organ recipients require long-term immunosuppression therapy along with frequent surveillance of the transplanted graft for indications of rejection, injury or failure. Long-term death rates in liver transplantation are more often attributable to long-term intake of immunosuppression medications than to liver graft dysfunction. Excessive immunosuppression can lead to declining kidney function, recurrent infections and other issues especially in the aging recipient population while suboptimal immunosuppression can lead to allograft injury, rejection or failure.

Monitoring for graft health post-transplant typically relies upon measurements of immunosuppression drug levels, serum liver enzyme testing, clinical symptoms of graft rejection and invasive liver biopsies. The measurement of serum liver enzymes may not reflect the full story as these enzymes are insensitive for predicting immune response and are considered to be late indicators of organ injury and/or damage given that by the time the enzymes are elevated the liver damage may have already occurred.

Currently, the gold standard for the detection of subclinical (before definitive, observable symptoms) graft injury is an invasive liver biopsy. Many times liver grafts will have abnormal histological findings late after transplantation despite having normal liver enzymes. Also, interpretation may be difficult in the presence of infection or recurrence of primary disease. As discussed, standard liver enzyme blood tests are non-specific and have an insensitivity for detecting subclinical graft injury. There is a need for non-invasive biomarkers to predict the onset and severity of rejection and improvement in histological markers to make an accurate diagnosis.

The identification of non-invasive biomarkers for subclinical graft injury to help individualize immunosuppression therapy especially in patients with autoimmune liver diseases will allow for better management of allograft protection along with improved management of adverse side effects. In this study, non-invasive biomarker assessment will be performed, utilizing TruGraf liver gene expression testing, to serially monitor for early immune activation prior to acute rejection with the aim to inform immunosuppression therapy management in liver transplant recipients with autoimmune diseases of the liver.

Primary Hypothesis Can utilization of Trugraf Liver gene expression testing to alter immunosuppression (IS) protocols in liver transplant recipients with autoimmune disease reduce the need for post-transplant liver biopsy as well as 1-year graft rejection rates as compared to a matched historical control group?

ELIGIBILITY:
Inclusion Criteria:

* Recipients ≥18 years of age
* Currently waitlisted for liver transplant or recipient of liver transplant within the last 30 days
* Primary indication for transplant due to autoimmune hepatitis (AIH) - Primary Biliary Cirrhosis (PBC) or Primary Sclerosing Cholangitis (PSC) etiologies
* First time, single-organ liver transplant recipient
* Willing and able to undergo protocol required TruGraf serial blood draws

Exclusion Criteria:

* Recipient <18 years of age
* Recipients of multi-organ or repeat transplantation
* Grafts from donors with HIV
* Grafts from donors with viremic Hepatitis A, B, C
* Inability to meet study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be recruited from the patient population of the Washington University liver transplant surgeons. These patients are routinely evaluated pre- and post- transplant by transplant surgeons. Patients who are on the waitlist for liver transplantation will be screened to determine if they meet the study eligibility criteria. Screening may occur either pre-transplant or post-transplant.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Graft survival | 12 months
  Organ recipients require long-term immunosuppression therapy along with frequent surveillance of the transplanted graft for indications of rejection, injury or failure.
Biopsy-Proven Acute Rejection (BPAR) results | 12 months
  Will be assessed via biopsy
Confirmed rejection diagnosis | 12 months
  Based on clinical data including the patient's symptoms and signs and confirmed by laboratory studies of blood and a tissue biopsy.
Clinical treatment of rejection | 12 months
  Possible revision to immunosuppressive (IS) medications

SECONDARY OUTCOMES:
Number of changes to immunosuppressive (IS) agents | 12 months
  Based on results of TruGraf liver gene expression test
Number of IS medications | 12 months
  % of patients achieving monotherapy immunosuppression
Immunosuppression reduction | 12 months
  % reduction from baseline
Estimated Glomerular filtration rate (eGFR) | 12 months
  eGFR change from baseline to month 12
Immune mediated issues | 12 months
  Infection incidence

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wellen, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University and Barnes Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri